CLINICAL TRIAL: NCT05039151
Title: Interstitial Fluid Composition in Patients With Septic Versus Non-septic Shock: an Exploratory Pilot Study
Acronym: INTERSEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LABRUYERE CRBFC-A 2020
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Liquid; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- septic shock: 50 patients with a diagnosis of septic shock established within 24 hours of admission with oedemas
  Interventions: Biological: interstitial fluid sampling; Biological: blood sampling
- control: 35 non-septic patients with oedema from another cause
  Interventions: Biological: interstitial fluid sampling; Biological: blood sampling

INTERVENTIONS:
Biological: interstitial fluid sampling — The sample will be taken via three small catheters (thinner than the catheters used for conventional infusions) under the skin in the abdomen. 1 to 10 ml of interstitial liquid will be collected. A sample will be taken on D1 and D2.
Biological: blood sampling — A blood sample (3 x 5 ml EDTA tubes) will be taken simultaneously. A sample will be taken on D1 and D2

SUMMARY:
Septic shock is a common reason for admission to intensive care units and severe infections are responsible for 6 million deaths a year worldwide. Fluid management appears to be a major issue in resuscitation and particularly in septic shock, where generalised oedema is almost systematic and is a major factor in poor prognosis during sepsis. The formation of oedema corresponds to an imbalance, according to Frank-Starling's law of the heart, between the vascular compartment and the interstitial compartment, which is composed of the interstitial liquid and an extracellular matrix. This extracellular matrix consists essentially of a network of collagen and fibroblast fibres. Even though all of the plasma in the body transits through the interstitium in 24 hours and desite its major importance in the microenvironment and intercellular communication, the interstitial compartment has not been fully described. In oncology, interstitial tissue seems to contribute to tumour growth through changes in matrix composition and pressure in the interstitium. This pressure actively contributes to the regulation of transcapillary filtration, and thus to the oedema and hypovolemia observed during sepsis. In usual conditions, the fibroblasts exert a tension on the collagen fibres of the matrix via integrin Beta-1 (ITGB1). This tension is released under the action of pro-inflammatory mediators, resulting in negative pressure which potentiates the formation of oedema.

It has been shown in an endotoxemia model that there is a thousandfold higher concentration of ITGB1 in the interstitium compared to the vascular compartment, suggesting a local secretion of this cytokine. The alteration of the extracellular matrix could also play a role in the perpetuation of oedema during septic shock. Considered as an organ in its own right, interstitial tissue is far from playing a passive role between the vascular compartment and the cells. The hypothesis is that interstitial fluid analysis could improve our understanding of the physiopathology of sepsis, in particular on the alteration of the mechanisms of fluid movement regulation, which remains very poorly understood while being closely associated with prognosis in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

COMMON INCLUSION CRITERIA

* Patient under mechanical ventilation and sedation
* Patient and/or trusted person (health care proxy) or close relative who has given their oral consent after being informed,
* Age ≥ 18 years old,

INCLUSION CRITERIA FOR THE SEPTIC SHOCK GROUP

* Diagnosis within 24 hours of admission of septic shock as defined by :
* A probable or confirmed infection
* And a SOFA score ≥ 2
* And the need to introduce vasopressors to obtain a MAP ≥ 65 mmHg despite adequate vascular filling
* And an arterial lactate > 2 mmol/l
* Norepinephrine dose greater than 0.1 μg/kg/min
* Septic shock present for less than 48 hours

INCLUSION CRITERIA FOR THE CONTROL GROUP

- Absence of sepsis and shock from any cause within 2 months prior to inclusion

Exclusion Criteria:

* Disseminated intravascular coagulation (DIC) with haemorrhagic syndrome
* Acute condition that can mimic sepsis :
* Acute pancreatitis without signs of superinfection
* Metformin Intoxication
* Patient with an unfavourable prognosis within 24 hours
* Patient under legal protection (safeguard of justice, guardianship or tutelage)
* Pregnant or breastfeeding women
* Patient not affiliated to national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ligible patients will be identified among patients admitted to Intensive Care Medicine
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
concentration of the differents components of the extracellular matrix on interstitial liquid at Day 1 | on Day 1
  Composition of the extracellular matrix on interstitial liquid on Day 1 (day of the first sampling) for the :
  * Type(s) of collagen by ELISA technique on 5L of liquid
  * Identification and quantification of interstitial glycosaminoglycans

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France